CLINICAL TRIAL: NCT05265364
Title: Acute and Late Toxicity After Moderate Hypo-fractionated Intensity Modulated Radiotherapy (IMRT) With Simultaneous Integrated Boost (SIB) for Prostate Cancer
Brief Title: Acute Toxicity After Moderate Hypo-fractionated Intensity Modulated Radiotherapy IMRT or Prostate Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: hanan fawzy (Other)
Responsible Party: Sponsor-Investigator, hanan fawzy, specialist of clinical oncology and nuclear medicin, Mansoura University Hospital
Organization: Mansoura University Hospital (Other)
Other Study IDs: MansouraUH
Record Dates: First submitted 2022-01-31; First posted 2022-03-03 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Radiation Toxicity
MeSH Terms: conditions — Radiation Injuries | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: IMRT with SIB — moderate hypofractioation using 2.5gy/fr in prostate cancer patients usig IMRT SIB technique

SUMMARY:
External radiation techniques (EBRT) is considered one of the primary therapies for patients of all risk classifications of prostate cacer . EBRT aims to control tumor growth while keeping acute and late adverse events to a minimum and ensuring biochemical progression-free outcome

DETAILED DESCRIPTION:
Patients and methods This is a prospective study of at least 50 patients to record acute and late toxicity using moderate hypo-fractionation with simultaneous integrated boost (SIB) IMRT for Prostate Cancer.Data will be collected at Clinical Oncology and Nuclear Medicine Department Mansoura University and Oncology Center Tanta University from January 2022 to December 2024 Patients Eligibility criteria Age >40 Pathologically proved prostate cancer Patients with unfavorable intermediate, High. very high risk groups and N1disease (Metastases in regional node(s) Risk groups according to NCCN guidelines 2021 and new grade grouping system of International Society of Urological Pathology (ISUP) Consensus Conference 2014

Unfavorable intermediate risk group :

exclusion criteria: Patients with prior pelvic irradiation. history of collagen vascular . inflammatory bowel disease. Double malignancy.

Methods Data acquisition planning computed tomography (CT) imaging will be performed in supine position using knee and ankle fixation support system for immobilization of the legs and patients arms on their chest.

Axial images will be obtained with 3-5 mm slice thickness from L1 vertebra to about 3 cm below the ischial tuberosity.

Before planning CT, patients will be instructed to have moderately, comfortably filled bladder and empty rectum four tattoos will be marked on the skin at the time of planning CT, rectum, bladder and hip joints will be contoured as organs at risk (OARs).

Target volumes

The prostate clinical target volume (CTV-pros) :

Include the whole prostate gland.

Prostate and seminal vesicles CTV (CTV-psv) :

Generated by 5mm expansion of CTV-pros in all directions except posteriorly at the prostate-rectum interface + proximal 2 cm of the seminal ( in case of cT3b the entire seminal vesicles will be included) .

Whole pelvis clinical target volume (CTV-pelv):

Consist of CTV-psv + common iliac (under L5-S1 space), external iliac, presacral and obturator lymph nodes.

Dose and fractionation All patients will receive moderate hypo fractionation with step and shoot IMRT with SIB in 28 fractions using 6-10 MV photon beams they will receive 70 Gy to PTV-pros in 2.5Gy/fraction and 57.4 Gy to PTV-psv in 2.05 Gy/fraction 50.4 Gy to the pelvic lymph nodes using 1.8 Gy/fraction for PTV coverage, the 95% of the prescribed dose will cover 95% of the target volume (V95% > 95%) for all PTVs. Rectum V45Gy, V63Gy, bladder V45Gy, hip joints V45Gy will be constrained below 50%, 20%, 65% and 10% of their volumes respectively.

Treatment delivery and care Before treatment a detailed medical history will be recorded and physical examination including PSA , pretreatment bone scan and pelvi -abdominal CT +/- MRI will be required to stage the prostate cancer and to exclude distant metastases.

Intermediate risk patients with bulky disease or un- favorable histological parameters will receive neo-adjuvant and concomitant hormone for 4-6 months (short-term hormone therapy) and in high risk patients neo-adjuvant ,concomitant and adjuvant hormone therapy for 24-36 months (long-term hormone therapy).

Patients will be evaluated every second week during the treatment, every three months after radiation therapy for the first year .

Acute toxicities will be reported during radiation therapy and within the initial 3-month and late toxicity will be recorded thereafter according to Common Terminology Criteria for Adverse Events (CTCAE)version 5.0 .

ELIGIBILITY:
Inclusion Criteria:

- Age >40 Pathologically proved prostate cancer Patients with unfavorable intermediate, High. very high risk groups and N1disease (Metastases in regional node(s)

Exclusion Criteria:

Patients with prior pelvic irradiation. history of collagen vascular . inflammatory bowel disease. Double malignancy.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male
Study Population: male patients with prostate cancer proved pathologically non metastatic
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-07-25 (Actual); Primary Completion 2024-12-12 (Estimated); Study Completion 2024-12-12 (Estimated)

PRIMARY OUTCOMES:
Primary end point is to asses acute toxicity of moderate hypo-fractionation using intensity-modulated radiotherapy (IMRT) with a simultaneous integrated boost (SIB) in prostate cancer patients | Acute toxicities will be reported within the initial 18 week of starting radiotherapy
  according to Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.

SECONDARY OUTCOMES:
Secondary end point is to asses late toxicity | will be recorded after 3 months of end of radiotherapy according to Common Terminology Criteria for Adverse Events (CTCAE)version 5.0 .
  using Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: hanan fawzy, Principal Investigator — Mansoura University Hospital
Locations (1):
- Clinical Oncology and Nuclear Medicin Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No